CLINICAL TRIAL: NCT02796729
Title: Detection of Metastatic Brain Tumours Using Dynamic Glucose Enhanced MRI After D-glucose Injection
Brief Title: CEST- Glucose Enhanced MRI for Metastatic Brain Tumours
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough enrollment
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Michael McKenzie, Radiation Oncologist, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H16-00646
Record Dates: First submitted 2016-06-01; First posted 2016-06-13 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Brain Neoplasms, Malignant; Metastasis
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Magnetic Resonance Spectroscopy; gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dynamic glucose enhanced MRI after D-glucose injection (Experimental): IV catheter preparation: Catheter will be placed in one arm. Fasting glucose levels measured with a glucometer using a 1-2 mL sample of blood. Only participants with normal fasting blood glucose levels (70-125 mg/dL) will proceed with the study. First IV catheter will monitor blood glucose every 10 min after bolus injection until it returns to normal. Second IV catheter is placed on the opposite arm for glucose infusion and GBCA (gadobutrol) infusion.
  Glucose infusion protocol: Occurs when the participant is in the MRI. Bolus injection of hospital grade 25g of 50% dextrose solution over 1 min is to increase blood glucose concentrations to about 3-4 times the normal level. Blood glucose levels should return to normal levels within 30 to 60 min.
  GBCA infusion protocol: Occurs when the participant is in the MRI; approximately 20 min after glucose infusion. Standard intravenous bolus injection of 0.1mM/kg of gadobutrol (Gadovist) at an injection rate of 5 mL/sec.
  Interventions: Procedure: Magnetic resonance imaging; Drug: Gadovist (Gadobutrol); Drug: 50% dextrose solution

INTERVENTIONS:
Procedure: Magnetic resonance imaging — MRI offers excellent images of the brain and is an important tool for diagnosing metastatic brain tumors. MRI scans are often used to plan treatments such as surgery and radiotherapy. When imaging participants with metastatic brain tumors, a contrast agent is often injected intravenously to highlight the relatively small tumours in the MRI. The standard metal-based MRI contrast agent is Health Canada approved and contains a material called gadolinium. MRI studies that use gadolinium-based contrast agents are called gadolinium enhanced MRI.
Drug: Gadovist (Gadobutrol) — Gadobutrol (INN) (Gd-DO3A-butrol) is a gadolinium-based MRI contrast agent (GBCA).
Drug: 50% dextrose solution — 50% Dextrose Injection, USP is a sterile, nonpyrogenic, hypertonic solution of dextrose in water for intravenous injection.

SUMMARY:
This project will compare two MRI contrast agents in metastatic brain tumours in humans. More specifically, the investigators will compare the tumour contrast obtained using glucose versus the current standard gadolinium-based contrast agent (GBCA, gadobutrol, trade name Gadovist, will be used).

First, participants will receive a glucose bolus injection followed by glucose enhanced MRI. Second, participants will receive a Gd-DTPA bolus injection followed by Gd-DTPA enhanced MRI. Both contrast studies will be performed during the same MRI study, which will be under one hour long.

DETAILED DESCRIPTION:
Purpose: To quantitatively compare glucose-enhanced MRI with the current standard GBCA enhanced MRI in participants with metastatic brain tumours prior to receiving radiotherapy from British Columbia Cancer Agency at Vancouver Cancer Centre.

Hypotheses: 1) Glucose enhanced MRI will highlight malignant metastatic brain tumours with comparable contrast to noise compared to GBCA and 2) Glucose enhancements in brain tumours will offer unique and complementary information, when compared to GBCA enhanced MRIs.

Justification: The current standard MRI contrast agent for metastatic brain tumours, GBCA, is limited by low specificity since GBCA accumulates in regions with disrupted blood brain barrier due to cancer as well as radiation necrosis and pseudo-progression after radiotherapy. It is important for radiation oncologists to reliably identify recurrent cancer, necrosis and post-treatment inflammation; and GBCA does not allow this. Therefore, a clinical need exists for an MRI technique that offers improved specificity for characterization of metastatic brain tumours before and after therapy. Glucose enhanced MRI represents a new technique that could offer improved specificity for detecting metastatic brain tumours.

Justification for number of participants included: The magnitude of signal enhancement is expected to vary between participants because 1) metastatic brain tumours exhibit a variety of enhancements patterns including ring, solid and nodular and 2) metastatic brain tumours will range in size. Therefore, 20 participants is considered sufficient to provide a reasonably accurate estimation of the expected mean tumour contrast as well as the expected variance in tumour contrast for future clinical trials. One additional healthy participant will be included in the study to perform a 'test-run' for the complicated MRI and infusion protocol.

Objectives:

1. Compare area under curve (AUC) maps calculated with glucose and GBCA in tumour and contralateral brain areas over different time intervals.
2. Compare post-injection contrast enhanced MRIs displaying maximum tumour contrast for single images to compare the 'instantaneous' contrast from both glucose enhanced and GBCA enhanced MRI.

Research Design and Statistical Analysis:

Participant recruitment: Recruitment will begin with collaborating radiation oncologists asking suitable patients if they are interested in participating in a MRI research study. The study will be described and if patients are still interested, consent will be taken and the screening forms will be completed. Participants will be scheduled for routine blood work to screen for eligibility (blood glucose status and renal function). Participants will also be scheduled for an MRI appointment at UBC MRI research centre.

Participants will be asked to fast the night before the MRI scan. They will be suggested to:"Eat a normal dinner and then not eat and only drink water from midnight until after the MRI scan, which will be scheduled in the morning to minimize the fasting duration."

MRI study details: To be performed at the UBC MRI research centre using a 3T Philips Achieva MRI.

Intravenous catheter preparation: Patients will arrive and an intravenous catheter will be placed in one arm by a qualified nurse or physician. Fasting glucose levels will be measured with a glucometer using a 1-2 mL sample of blood. Only participants with normal fasting blood glucose levels (70-125 mg/dL) will proceed with the study. The first intravenous catheter will be used to monitor blood glucose every 10 minutes after bolus injection until it returns to normal. A second intravenous catheter is placed on the opposite arm for glucose infusion and GBCA (gadobutrol) infusion.

Glucose infusion protocol: This will occur when the participant is lying in the MRI. The protocol mimics the intravenous glucose tolerance test. Bolus injection of hospital grade 25g of 50% dextrose solution over 1 minute is used to increase blood glucose concentrations to approximately 3-4 times the normal level. Blood glucose levels should return to normal levels within 30 to 60 minutes according to previous studies.

GBCA infusion protocol: This will also occur when the participant is lying in the MRI and approximately 20 minutes after glucose infusion. Standard intravenous bolus injection of 0.1mM/kg of gadobutrol (Gadovist) at an injection rate of 5 mL/sec.

MRI timeline: Metastatic tumours will be initially detected using standard 3D T2-weighted MRI. Then a slice of interest containing maximum tumour coverage will be selected for the remainder of the study. In participants with multiple metastases, the largest untreated lesion will be the focus and multiple lesions will be included if feasible.

MRI scans will include: 1) Scouts and magnetic field shimming; 2) 3D T2 weighted MRI; 3) Magnetic field maps (B0 & B1); 4) Pre- glucose injection Z-spectrum; 5) Begin serial glucose enhanced MRI; [glucose infusion after 3 minutes]; 6) Post- glucose injection Z-spectrum after 10 minutes; 7) Begin serial T1-weighted gadobutrol enhanced MRI; [gadobutrol infusion after 3 minutes]; 8) Continue Gd-enhanced MRI scans until 10 minutes post-injection.

MRI data analysis will be performed using well documented, standard techniques using custom-built Matlab software.

Statistics: Mean and standard deviation statistics will be calculated for both glucose enhanced and gadobutrol enhanced data. Tumour contrast to noise will be calculated using AUC curves as well as single MR images. These metrics will help to quantify the tumour detection sensitivity of glucose enhanced MRI relative to GBCA enhanced MRI. The investigators expect that both techniques will offer similar contrast to noise in metastatic tumours, based on previously reported results in human participants with glioma tumours.

ELIGIBILITY:
Inclusion Criteria:

* Male or females
* Between 18 and 65 years of age
* Of all ethnic groups
* BCCA participants with at least one contrast enhancing brain mass with a diameter ≥ 1 cm and consistent with metastatic carcinoma*
* Able to give consent
* Willingness to participate in the study * One additional healthy participant will be included in the study to perform a 'test-run' for the complicated MRI and infusion protocol.

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus (self-reported or HbA1C ≥ 6.5%)
* Ferromagnetic implant or foreign metallic bodies (pacemaker, loose metal, etc.)
* Claustrophobia
* History of kidney disease and/or eGFR < 60
* Abnormal fasting blood glucose (<70mg/dL or >125 mg/dL)
* Allergic to corn
* History of adverse reactions to gadolinium based contrast agents
* Poor performance status (Karnofsky PS<70%)
* Previously received whole brain radiotherapy
* All lesions evident on imaging were previously treated with stereotactic radiosurgery
* The participants weigh more than 300lbs
* The participants had surgery in the last 6 weeks
* The participants have an intrauterine device
* The participants have cosmetic tattoos

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Integral tumour contrast generated by GBCA and glucose experiments will be assessed using Area Under Curve (AUC). | 1h procedure
  Area Under Curve (AUC) is measured using a sequence of MR images acquired before and after contrast injection. AUC values will be compared in tumour and contralateral brain areas to calculate the integral tumour contrast generated by glucose and GBCA experiments.

SECONDARY OUTCOMES:
Maximum instantaneous tumour contrast generated by GBCA and glucose experiments will be assessed. | 1h procedure
  This metric is calculated using a single MR image acquired before contrast injection and a single image acquired after injection. The pair of images (before and after) that generates the maximum contrast is used. This metric will be used to compare contrasts generated by glucose and GBCA experiments.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McKenzie, Principal Investigator — BCCA
Locations (1):
- BC Cancer Agency- Vancouver Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Only participants (and their most responsible physician with permission) have the option of receiving their own personal data.

REFERENCES:
- [Background] Chan KW, McMahon MT, Kato Y, Liu G, Bulte JW, Bhujwalla ZM, Artemov D, van Zijl PC. Natural D-glucose as a biodegradable MRI contrast agent for detecting cancer. Magn Reson Med. 2012 Dec;68(6):1764-73. doi: 10.1002/mrm.24520. Epub 2012 Oct 16. PMID 23074027
- [Background] Nasrallah FA, Pages G, Kuchel PW, Golay X, Chuang KH. Imaging brain deoxyglucose uptake and metabolism by glucoCEST MRI. J Cereb Blood Flow Metab. 2013 Aug;33(8):1270-8. doi: 10.1038/jcbfm.2013.79. Epub 2013 May 15. PMID 23673434
- [Background] Walker-Samuel S, Ramasawmy R, Torrealdea F, Rega M, Rajkumar V, Johnson SP, Richardson S, Goncalves M, Parkes HG, Arstad E, Thomas DL, Pedley RB, Lythgoe MF, Golay X. In vivo imaging of glucose uptake and metabolism in tumors. Nat Med. 2013 Aug;19(8):1067-72. doi: 10.1038/nm.3252. Epub 2013 Jul 7. PMID 23832090